CLINICAL TRIAL: NCT03053622
Title: A Phase 1, Single-Dose Study to Assess the Relative Bioavailability, Absolute Bioavailability, and Tolerability of LY3074828 Formulations in Healthy Subjects
Brief Title: A Study of Mirikizumab (LY3074828) Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16542; I6T-MC-AMAL (Other: Eli Lilly and Company); 2016-003584-18 (EudraCT Number)
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mirikizumab Test Subcutaneous (SC) 1 (Experimental): 250 mg mirikizumab test formulation given as a single injection SC in healthy participants
  Interventions: Biological: Mirikizumab Test
- Mirikizumab Test SC 2 (Experimental): 250 mg mirikizumab test formulation given as two injections given SC in healthy participants
  Interventions: Biological: Mirikizumab Test
- Mirikizumab Test Intravenous (IV) (Experimental): 250 mg mirikizumab test formulation given as an infusion into the vein in healthy participants
  Interventions: Biological: Mirikizumab Test
- Mirikizumab Reference (Active Comparator): 250 mg mirikizumab reference formulation given as three injections subcutaneous (SC) in healthy participants
  Interventions: Biological: Mirikizumab Reference

INTERVENTIONS:
Biological: Mirikizumab Test — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab Test SC 2; Mirikizumab Test Subcutaneous (SC) 1
Biological: Mirikizumab Test — Administered IV
  Other Names: LY3074828
  Arms: Mirikizumab Test Intravenous (IV)
Biological: Mirikizumab Reference — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab Reference

SUMMARY:
This study is conducted to compare how much mirikizumab, in two different formulations, is absorbed into the bloodstream and how long the body takes to get rid of it, when given as an injection under the skin or into the veins. Side effects of the injection will be collected. Each participant will be in the study for about 18 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a screening body mass index (BMI) of greater than 18 and less than or equal to 32 kilograms per meter squared (kg/m²), inclusive
* Have medical test results that are acceptable for the study
* Must be willing to make oneself available for the whole study and be willing to follow study procedures

Exclusion Criteria:

* Are currently participating or recently participated in a clinical trial or any other type of medical research judged to be incompatible with this study
* Have known allergies to compounds or drugs similar to Mirikizumab
* Have previously participated or withdrawn from this study
* Have or used to have health problems or medical test results that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirikizumab Test SC 1: 250 mg mirikizumab test formulation given as a single injection SC in healthy participants
Period: Overall Study
Arm/Group | Mirikizumab Reference | Mirikizumab Test SC 2 | Mirikizumab Test SC 1 | Mirikizumab Test Intravenous (IV)
Started | 17 | 16 | 17 | 17
Received at Least One Dose of Study Drug | 17 | 16 | 17 | 17
Completed | 17 | 16 | 17 | 16
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirikizumab Reference | Mirikizumab Test SC 2 | Mirikizumab Test SC 1 | Mirikizumab Test Intravenous (IV) | Total
Number analyzed (Participants) | 17 | 16 | 17 | 17 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.3) | 40.7 (18.0) | 52.1 (9.6) | 43.6 (14.9) | 45.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 9 | 8 | 28
  Male | 11 | 11 | 8 | 9 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 17 | 16 | 17 | 15 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 3
  White | 17 | 13 | 17 | 16 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 17 | 16 | 17 | 17 | 67

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From 0 to Infinity (AUC[0-∞]) of Mirikizumab
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from 0 to Infinity (AUC[0-∞]) of Mirikizumab
Time Frame: 0,end of infusion,2,6 hours(h); 24 h; 72 h; 168 h; 240 h; 336 h; 504 h; 672 h; 1008 h; 1344 h; 1680 h; 2016 h, post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram* Day/Milliliter(µg*day/mL)
Arm/Group | Mirikizumab Reference | Mirikizumab Test SC 2 | Mirikizumab Test SC 1 | Mirikizumab Test Intravenous (IV)
Number analyzed (Participants) | 17 | 16 | 17 | 17
Microgram* Day/Milliliter(µg*day/mL) | 215 (31) | 214 (55) | 293 (36) | 695 (22)
Statistical Analysis 1: Comparison: Mirikizumab Reference vs Mirikizumab Test SC 2; Test type: Other; Ratio of Geometric Least Squares Means = 0.996, 90% CI 2-sided [0.807 to 1.23]
Statistical Analysis 2: Comparison: Mirikizumab Test SC 2 vs Mirikizumab Test SC 1; Test type: Other; Ratio of Geometric Least Squares Means = 0.729, 90% CI 2-sided [0.591 to 0.898]
Statistical Analysis 3: Comparison: Mirikizumab Test SC 1 vs Mirikizumab Test Intravenous (IV); Test type: Other; Ratio of Geometric Least Squares Means = 0.422, 90% CI 2-sided [0.343 to 0.518]
Statistical Analysis 4: Comparison: Mirikizumab Test SC 2 vs Mirikizumab Test Intravenous (IV); Test type: Other; Ratio of Geometric Least Squares Means = 0.307, 90% CI 2-sided [0.249 to 0.379]

2. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Mirikizumab
Description: PK: Maximum Observed Concentration (Cmax) of Mirikizumab
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/Milliliter (µg/mL)
Arm/Group | Mirikizumab Reference | Mirikizumab Test SC 2 | Mirikizumab Test SC 1 | Mirikizumab Test Intravenous (IV)
Number analyzed (Participants) | 17 | 16 | 17 | 17
Microgram/Milliliter (µg/mL) | 11.4 (34) | 11.2 (51) | 14.9 (32) | 90.0 (14)
Statistical Analysis 1: Comparison: Mirikizumab Reference vs Mirikizumab Test SC 2; Test type: Other; Ratio of Geometric Least Squares Means = 0.986, 90% CI 2-sided [0.810 to 1.20]
Statistical Analysis 2: Comparison: Mirikizumab Test SC 2 vs Mirikizumab Test SC 1; Test type: Other; Ratio of Geometric Least Squares Means = 0.753, 90% CI 2-sided [0.619 to 0.916]

3. Secondary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Mirikizumab
Description: PK: Time of Maximum Observed Drug Concentration (Tmax) of Mirikizumab
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Mirikizumab Reference | Mirikizumab Test SC 2 | Mirikizumab Test SC 1 | Mirikizumab Test Intravenous (IV)
Number analyzed (Participants) | 17 | 16 | 17 | 17
Hour (h) | 73.12 [72.45 to 145.82] | 73.41 [72.67 to 240.67] | 73.25 [72.22 to 145.30] | 2.00 [0.50 to 2.15]
Statistical Analysis 1: Comparison: Mirikizumab Reference vs Mirikizumab Test SC 2; Test type: Other; Median Difference (Final Values) = 0.28, 90% CI 2-sided [-0.10 to 48.40]
Statistical Analysis 2: Comparison: Mirikizumab Test SC 2 vs Mirikizumab Test SC 1; Test type: Other; Median Difference (Final Values) = 0.25, 90% CI 2-sided [-0.25 to 23.97] — In this outcome, the median difference is not calculated by subtracting two observations, it is derived by "Hodges-Lehmann approach to estimating location shift". This method will give the value of 0.25

ADVERSE EVENTS:
Time Frame: Up To 4 Months
Description: All participants who received at least one dose of study drug.
Arm/Group | Mirikizumab Reference | Mirikizumab Test SC 2 | Mirikizumab Test SC 1 | Mirikizumab Test Intravenous (IV)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 17/17 | 15/16 | 17/17 | 15/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirikizumab Reference (N=17) | Mirikizumab Test SC 2 (N=16) | Mirikizumab Test SC 1 (N=17) | Mirikizumab Test Intravenous (IV) (N=17)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 17 (47) | 15 (33) | 17 (18) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 2 (2) | 1 (1) | 7 (7)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (7)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bladder irritation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03053622/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03053622/SAP_001.pdf